CLINICAL TRIAL: NCT05812638
Title: Effects of Mental Imagery With Virtual Reality Training on Lower Limb Functions in Stroke
Brief Title: Mental Imagery for Lower Limb Functions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01261 Tasmiya
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Imagery (Experimental): For mental imagery, the calm and nice atmosphere isrequired for the patientsto focus on the details while sitting on a chair. The audiotape and headphones are given to the patients. The audiotape tape comprised of three phases. The first phase is relaxation phase. The patient has to do the first phase actively. In this phase patients have asked to do the deep breathing exercises while sitting on a chair and then contract their lower limb muscles from distal to proximal. The second phase is task-oriented phase. The patient has to imagine him performing the tasks.
  Interventions: Other: Mental imagery technique
- Virtual Reality (Active Comparator): The virtual reality training will be given through Kinect connected with Xbox 360.
  The Xbox games used are 20,000 water leaks, reflex ridge and river rush. The spacious environment will be given and walker are sometimes required for assistance. The LED and system are 3 feet away from patients. The VR training will be given to the both control and experimental groups
  Interventions: Other: Virtual Reality technique

INTERVENTIONS:
Other: Mental imagery technique — Warm up Period Mental Imagery (Sit-stand task Static stance (30 seconds) Indoor walk on a leveled surface Walk indoor towards target Forward / Side Stepping) Walk outdoors
  Arms: Mental Imagery
Other: Virtual Reality technique — Virtual reality training (River rush, 20000 water leaks, reflex ridge.)
  Arms: Virtual Reality

SUMMARY:
Stroke is a neurological impairment occurs due to cardiovascular abnormality and cerebrovascular disease. The term 'stroke' is mostly used when there is sudden loss of function of the body due any abrupt changes.The rates of disability are increasing along with mortality and morbidity rates due to stroke. The poor motor performance of lower limb affects gait severely. The slow velocity and other gait deviations limit the stroke survivors' ability to perform ADL's and interfere with their quality of life.

Hence, rehabilitation is obligatory for these patients to improve their quality of life

DETAILED DESCRIPTION:
motor imagery is helpful in improving mobility in healthy and neurologically impaired patients. When the patient is asked to do a movement, for example the patient is asked to walk along a draw line and then that patient has to imagine this same action in kinesthetic imagery. Neuroimaging shows that brain areas are more or less activated in the same manner. It can be concluded that there is some relation between mental imagery ability and muscular actions. In the stroke patients who have intact ability of mental imagery show activation of cortical areas demonstrating its ability to activate sub cortical areas also. Therefore, these results amplify the concept of using mental imagery for rehabilitation purpose of even deep lesion in motor nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients (both genders)
* Age 40-60 years
* Patients with sub-acute/ chronic stroke (>3 months)
* Modified Ashworth Ranking Scale 1-3
* MOCA scoring >24-30

Exclusion Criteria:

* Any active pathological condition
* Visual or hearing impairment
* Orthopedic issues hindering Mobility Substantially (Fractures, Severe Degenerative
* Joint Diseases etc.)
* Psychological issues

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Assessment Scale - Lower Extremity | week 6
  This scale is recognized as a golden standard for assessment of motor function of stroke patients worldwide. It focuses on reflex activity, voluntary movements within and outside of synergies, ability to perform isolated movement, and coordination
Berg Balance Scale | week 6
  In elderly Population, BBS is most commonly used outcome measure for functional balance. It is 14 Item balance measure scored on 5-point ordinal scale with range of 0 to 4, where high score indicates good balance & decreased risk of fall and vice versa.
  A maximum score of 56 is achievable
Timed Up and Go test | week 6
  It is used to assess functional mobility; the risk of fall and dynamic balance can also be determined. In TUG test, the participant is asked to get up from a chair, walk a distance of 3 meters at Regular pace, turn around, walk a distance of 3 meter back to the chair and sit down
10-meter walk test | week 6
  In this test, the participant walks through a 10-m walkway without any break. At the 4- m of walkway, time is recorded in order to obtain a rhythmic phase of walking speed
Wisconsin Gait Scale | week 6
  This scale is used to assess gait cycle. It consists of 14 items, the higher the score, greater will be the disability. These scale focuses on the components of stance phase, guardedness of affected leg, toe off, swing phase and heel strike

CONTACTS AND LOCATIONS:
Overall Officials: arshad Malik, Phd, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No